CLINICAL TRIAL: NCT03410342
Title: The Effects of Types of Fruits and Vegetables on Vascular Function in Prehypertensive Participants: a Pilot Study
Brief Title: The Effects of Types of Fruits and Vegetables on Vascular Function
Acronym: CIRCUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: Imperial College London (Other)
Responsible Party: Principal Investigator, Linda Oude Griep, Senior Research Associate, University of Cambridge
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 17HH3878; Research Ethics Committee (Registry Identifier: 17/LO/0862)
Record Dates: First submitted 2017-12-03; First posted 2018-01-25 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Blood Pressure; Vascular Stiffness; Cardiovascular Risk Factor
Keywords: Blood Pressure; Vascular Stiffness; Cardiovascular Risk Factor; Fruit and vegetable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Fruits and Vegetables (LFV) (Placebo Comparator): 1 portion of fruits plus 1 portion of vegetables, of commonly consumed types per day.
  Intakes are at 25th percentile of UK consumption (NDNS) and will exclude citrus fruits, cruciferous and allium vegetables.
  Interventions: Other: LFV
- High Fruits and Vegetables (HFV) (Experimental): 4 portions of fruits plus 4 portions of vegetables, of commonly consumed types per day excluding citrus fruits, cruciferous and allium vegetables.
  Interventions: Other: HFV
- High Citrus fruits and Cruciferous vegetables (CC) (Experimental): 4 portions of citrus fruits plus 4 portions of cruciferous vegetables per day excluding any other types of fruits and vegetables including allium vegetables.
  Interventions: Other: CC

INTERVENTIONS:
Other: LFV — 1 apple/banana/small bunch of grapes per day plus 1 portion of carrot/pepper/tomato per day
  Arms: Low Fruits and Vegetables (LFV)
Other: HFV — 4 portions of fruits (apples, bananas, grapes, pears) plus 4 portions of vegetables (carrots, cucumber, sweet peppers, tomatoes), of commonly consumed types per day excluding citrus fruits, cruciferous and allium vegetables.
  Arms: High Fruits and Vegetables (HFV)
Other: CC — 4 portions of citrus fruits (clementines, grapefruits, lemons, oranges) plus 4 portions of cruciferous vegetables (broccoli, brussels sprouts, cauliflower, kale, savoy cabbage) per day.
  Arms: High Citrus fruits and Cruciferous vegetables (CC)

SUMMARY:
The CIRCUS study is a randomised controlled, cross-over trial to evaluate the effects of increased intakes of citrus fruits and cruciferous vegetables on vascular function in 36 untreated, prehypertensive participants.

DETAILED DESCRIPTION:
The study comprises three 14-day dietary intervention periods, preceded by one week run-in period and separated by one week wash-out periods, 9 weeks in total. The diet will be fully controlled and provided by the researchers. Participants will receive in random order three interventions:

* 1 portion of fruits plus 1 portion of vegetables, of commonly consumed types per day. Intakes are at 25th percentile of UK consumption and will exclude citrus fruits, cruciferous and allium vegetables.
* 4 portions of fruits plus 4 portions of vegetables, of commonly consumed types per day excluding citrus fruits, cruciferous and allium vegetables.
* 4 portions of citrus fruits plus 4 portions of cruciferous vegetables per day.

ELIGIBILITY:
Inclusion Criteria:

* 40 - 65 years
* Average systolic blood pressure of 125-140 mmHg at 2 measurements separated by >30 minutes
* No use of antihypertensive medication
* No reported current or previous diabetes mellitus, (secondary) hypertension, or metabolic, cardiovascular, renal, liver, thyroid, gastrointestinal diseases
* Body Mass Index between 20 - 35 kg/m2
* Non-smoker
* Average fruit and vegetable consumption of <4 portions per day (UK average, 40-65 years), or willing to reduce habitual daily fruit and vegetable intake.

Exclusion Criteria:

* Any medication likely to interfere with energy metabolism, appetite regulation and hormonal balance.
* Excessive alcohol intake of > 21 units per week (females) or >28 units per week (male) and not willing to limit alcohol intake to maximum of 1 unit/day
* Physical activity of >=10 hours/week of moderate to vigorous physical activity
* Weight loss or gain of >=3 kg in the preceding 3 months
* Use of dietary supplements or unwilling to stop supplement use >= 2 weeks before enrolment and during intervention
* Pregnancy or lactation
* Intervention specific factors, including:

  * Unable or unwilling to consume provided diets during the intervention
  * Unsufficient storage space for provided diets
  * Food sensitivities or vegetarian/vegan diet by choice
  * Participation in another intervention study at the same time
  * Living > 15 miles from the Imperial/NIHR Clinical Research Facility at Hammersmith Hospital
  * No signed informed consent

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-06-21 (Actual)

PRIMARY OUTCOMES:
Blood pressure | Measured on the morning after each of three recurring run-in periods and after each of three recurring 2-week intervention periods, 6 times total during 9 weeks
  Changes in systolic and diastolic blood pressure (mmHg) measured by automated oscillometric device (average of 3 measurements).

SECONDARY OUTCOMES:
Arterial stiffness | Measured on the morning after each of three recurring run-in periods and after each of three recurring 2-week intervention periods, 6 times total during 9 weeks
  Changes (end minus baseline values) in arterial stiffness (pulse wave analysis)
Markers of cardiometabolic health measured in fasted blood samples | Measured on the morning after each of three recurring run-in periods and after each of three recurring 2-week intervention periods, 6 times total during 9 weeks
  e.g. high-density lipoprotein
Markers of endothelial function measured in fasted blood samples | Measured on the morning after each of three recurring run-in periods and after each of three recurring 2-week intervention periods, 6 times total during 9 weeks
  e.g. C-Reactive Protein
Markers of low-grade inflammation measured in fasted blood samples | Measured on the morning after each of three recurring run-in periods and after each of three recurring 2-week intervention periods, 6 times total during 9 weeks
  e.g. Interleukin-6
Urinary metabolic profiles | Measured on the morning after each of three recurring run-in periods and after each of three recurring 2-week intervention periods, 6 times total during 9 weeks
  (Un)targeted metabolic profiling by NMR and MS
Circulatory metabolic profiles | Measured on the morning after each of three recurring run-in periods and after each of three recurring 2-week intervention periods, 6 times total during 9 weeks
  (Un)targeted metabolic profiling by NMR and MS
Established objective markers of food intake | Measured on the morning after each of three recurring run-in periods and after each of three recurring 2-week intervention periods, 6 times total during 9 weeks
  e.g. vitamin C
Faecal microbiome composition | Measured on the morning after each of three recurring run-in periods and after each of three recurring 2-week intervention periods, 6 times total during 9 weeks
  Measured by 16SrRNA gene sequencing
Cognitive function | Measured on the morning after each of three recurring run-in periods and after each of three recurring 2-week intervention periods, 6 times total during 9 weeks
  e.g. Stroop-test
Self-rated general health and mental well-being | Measured on the morning after each of three recurring run-in periods and after each of three recurring 2-week intervention periods, 6 times total during 9 weeks
  e.g. Positive and Negative Affect Schedule (PANAS) that consists of two 10-item scales to measure both positive and negative affect. Each item is rated on a Likert scale of 1 (not at all) to 5 (very much). Positive and negative affect scores are added seperately to a reange from 10 to 50. Higher positive scores represents higher levels of positive affect. Lower negative scores respresaent lower levels of negative affect.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Oude Griep, PhD, Principal Investigator — MRC Epidemiology Unit, University of Cambridge
Locations (2):
- United Kingdom (2):
  - Cambridge Epidemiology & Trials Unit, Cambridge
  - Imperial/NIHR Clinical Research Facility, London

IPD SHARING:
Plan to Share IPD: Yes
As describe in study protocol
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: In a timely manner when results have been published in peer-reviewed journals.

DOCUMENTS (2):
  • Study Protocol (2019-11-19): https://cdn.clinicaltrials.gov/large-docs/42/NCT03410342/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-04): https://cdn.clinicaltrials.gov/large-docs/42/NCT03410342/SAP_001.pdf